CLINICAL TRIAL: NCT01874223
Title: Prospective Validation of Cough, Dyspnea, and Quality of Life Questionnaires in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Prospective Validation of Cough, Dyspnea, and Quality of Life Questionnaires in Patients With IPF
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 23346
Record Dates: First submitted 2013-05-06; First posted 2013-06-10 (Estimated); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis
Keywords: Interstitial Lung Disease (ILD); Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IPF-diagnosed patients: A group of up to 40 patients with a diagnosis of mild to severe IPF per American Thoracic Society (ATS) guidelines, either with no cough at baseline to severe cough at baseline, will be followed for at least a one-time assessment and every six months for up to 18 months to establish validity, responsiveness, and reliability of cough, dyspnea, and QOL instruments in patients with IPF.

SUMMARY:
The purpose of this study is to test cough, dyspnea (shortness of breath), and quality of life (QOL) questionnaires for their accuracy, sensitivity, and ability to reliably measure the severity of cough, breathlessness, and changes in cough and disease-related quality of life over time in Idiopathic Pulmonary Fibrosis (IPF) patients. These questionnaires have been used in other types of disease, but have not all been tested and validated in patients with cough due to IPF. Our hypothesis is that worsening of cough, dyspnea, and cough-related QOL questionnaire scores will correlate with physiologic markers of IPF severity and worsening of disease. Written, valid questionnaires measuring cough, dyspnea, and QOL are important to assess the benefit of investigational drugs under development to treat patients with IPF.

DETAILED DESCRIPTION:
This study in patients with IPF will determine the validity, responsiveness, and reliability of two cough measures (the Leicester Cough Questionnaire (LCQ), as well as Visual Analogue Scales (VASs) for cough severity and distress; one dyspnea measure (the Baseline and Transition Dyspnea Index (BDI/TDI); and two health-related quality of life (HRQL) measures (the obstructive lung disease-specific Saint George's Respiratory Questionnaire (SGRQ) and the IPF-specific 'A Tool to Assess QOL in IPF' (ATAQ-IPF). Both the SGRQ and ATAQ include cough questions. Study participants will complete all questionnaires at baseline, 6, 12, and 18 months at the time of their usual clinic visits. Physiologic data will be collected at the same time of these visits including pulmonary function testing, exercise oxygen saturation, and changes in medications and health status. Changes in cough, dyspnea and QOL scores will be correlated with concurrent changes in physiologic markers of IPF severity. If a study participant has an acute worsening of their IPF, or undergoes lung transplantation, study questionnaires may be given at these additional timepoints when possible.

ELIGIBILITY:
Inclusion Criteria:

* Completion of informed consent.
* Adults over the age of 18.
* Diagnosis of IPF per ATS guidelines.
* Clinically stable at the time of enrollment defined as no antibiotics within the past month, with the exception of those patients currently listed for Lung Transplantation.
* No changes in immunosuppressive regimens (if applicable) over past month.

Exclusion Criteria:

* Inability to understand or complete paper and pencil questionnaires.
* Patient not planning to return to Stanford for clinic visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IPF as defined by ATS guidelines
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-11-04 (Actual)

PRIMARY OUTCOMES:
Correlation of LCQ scores with physiologic markers of IPF severity | Baseline, 6, 12 and 18 months
  Change scores for the LCQ cough-related quality of life instrument will be correlated with changes in pulmonary function tests

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mohabir, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Chest Clinic, Stanford, California, United States